CLINICAL TRIAL: NCT04282200
Title: The Use of Intravenous Ketorolac in a Multimodal Approach to Pain Management in Acute Pancreatitis
Brief Title: Ketorolac in Acute Pancreatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Anthony Gentene, Clinical Pharmacy Specialist, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0283
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (No Intervention): Patients receiving standard of care pain management including opioids.
- Ketorolac (Active Comparator): Patients will receive standard of care pain management plus intravenous ketorolac.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — intravenous ketorolac 30 mg every 6 hours
  Arms: Ketorolac

SUMMARY:
This study will compare pain management strategies for patients hospitalized with acute pancreatitis. Standard of care pain management will be compared to standard of care plus intravenous ketorolac.

DETAILED DESCRIPTION:
Patients hospitalized for acute pancreatitis and admitted to an internal medicine team will be eligible for study. Patients enrolled will be blindly randomized to receive open-label pain management of standard of care or standard of care plus intravenous ketorolac. Patients will be enrolled between hour 24 and 48 of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* opioid order for pain secondary to acute pancreatitis
* diagnosis of acute pancreatitis defined by the presence of two of the following three criteria: abdominal pain, lipase > 3x upper limit of normal, and/or findings of AP on imaging
* a patient with acute-on-chronic pancreatitis that does not exhibit elevated lipase levels is eligible for inclusion if the patient has the other two criteria
* received at least 3 L of IV crystalloid fluid within first 24 hours of admission to ensure patients have received initial volume expansion
* hemodynamically stable represented by a mean arterial blood pressure (MAP) of ≥65 mmHg
* female patients not documented in chart as post-menopause must have a negative pregnancy test

Exclusion Criteria:

* history of chronic heart failure
* history of acute coronary syndrome (ST-elevation myocardial infarction (STEMI) or non-ST elevation myocardial infarction (NSTEMI)) within last 6 months
* history of ischemic or hemorrhagic stroke within last 6 months
* history of upper gastrointestinal bleed (GI) within last 6 months
* history of inflammatory bowel disease
* history of cirrhosis
* any overt, active bleeding requiring blood transfusion
* considered to be high bleed risk (platelet < 50,000/mcL)
* pregnant or breastfeeding
* prisoners
* cognitively impaired patients: not alert and oriented to person, place, and time (patient must be able to consent)
* allergy to NSAIDs, ketorolac, or aspirin
* admission to an intensive care unit
* evidence of infected pancreatitis (i.e. abscess) on imaging studies
* acute kidney injury or chronic kidney disease with CrCl<30

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Opioid use during study enrollment | day 1 to day 5 of study
  oral morphine equivalents (OME)

SECONDARY OUTCOMES:
Day-to-day oral morphine equivalents | day 1 to day 5 of study
  Compare opioid use in each day of study
Duration of intravenous opioid use | During hospital admission
  compare duration of need for IV opioids and transition to oral opioids

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Gentene, PharmD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No